CLINICAL TRIAL: NCT05995769
Title: Mechanisms Supporting Psilocybin-assisted Psychotherapy for Alcohol Use Disorder: A Randomized, Controlled Clinical Trial
Brief Title: Psilocybin-Assisted Psychotherapy for Alcohol Use Disorder
Acronym: PAP-AUD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Johns Hopkins University (Other); University of Maryland (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB23-0666
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-08

CONDITIONS: Alcohol Use Disorder; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dose (25mg) (Experimental): PEX010 (Oral Psilocybin), 25mg; single dose administered 24hrs prior to first of 5 weekly MET sessions
  Interventions: Drug: Psilocybin
- Low dose (1mg) (Active Comparator): PEX010 (Oral Psilocybin), 1mg; single dose administered 24hrs prior to first of 5 weekly MET sessions
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Single dosing session followed by 5 MET weekly sessions starting 24hrs after dosing
  Other Names: magic mushrooms; PEX010

SUMMARY:
The aim of this study is to determine if a single dose of psilocybin administered with motivational enhancement therapy (MET) can reduce heavy drinking in patients with an alcohol use disorder (AUD).

DETAILED DESCRIPTION:
The primary objective of this study is to determine if psilocybin administered with a standardized psychotherapeutic intervention, motivational enhancement therapy (MET), can reduce heavy drinking in a patient population with an alcohol use disorder (AUD). Patients with an AUD will be randomly allocated to either a high dose (25mg; active treatment) or a low dose (1mg; active control) psilocybin arm. All participants will receive 5 sessions of MET, starting at 24hrs post-dosing. Heavy drinking will be assessed as percent heavy drinking days using the Time Line Follow Back (TLFB) at baseline and 1-, 4-, and 12-weeks post-dosing.

A total of 128 male and female patients between the ages of 22-65 with a moderate to severe AUD diagnosis will be recruited from the community. Participants will undergo a thorough screening procedure and eligible participants will be randomly allocated to the high (N=64) or low (N=64) psilocybin doses. All participants will complete a baseline session consisting of clinical, behavioral, and neuroimaging measures. Following the single dosing session, participants will complete 5 weekly MET sessions. Neuroimaging measures will be assessed again at 1-week post-doing. Clinical and behavioral outcomes will be measured at 1-, 4-, and 12-weeks post-dosing

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 AUD criteria of at least moderate severity
* Meets heavy drinking requirements (heavy drinking days, number of drinks) in past 30 days
* Desire to decrease alcohol consumption
* Limited lifetime hallucinogen use

Exclusion Criteria:

* Severe or moderate substance use disorder other than alcohol or nicotine in past 6 months
* Diagnosis of schizophrenia, bipolar disorders or first-degree relative with diagnosis
* Active suicidal ideation or serious attempt within past 3 years
* Currently pregnant, nursing, or trying to become pregnant
* Any notable abnormality on ECG, physical exam, or routine medical blood laboratory test

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Heavy drinking | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  Percent heavy drinking days (TLFB)

SECONDARY OUTCOMES:
Abstinence | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  Days abstinent (TLFB)
Biomarkers of alcohol consumption | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  Phosphatidylethanol (Peth)
Alcohol cue reactivity | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  Alcohol urge questionnaire (AUQ)
Cognitive flexibility | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  Berg Card Sorting Task
Depression | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  The Montgomery-Åsberg Depression Rating Scale (MADRS)
Anxiety | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  The General Anxiety Disorder 7 (GAD-7) scale
Quality of life | Change from baseline to 1-, 4-, and 12-weeks post-dosing
  The World Health Organization Quality of Life (WHOQOL) scale
Glutamate levels | Change from baseline to 1-week post-dosing
  MR spectroscopy of glutamate levels in the anterior cingulate cortex
GABA levels | Change from baseline to 1-week post-dosing
  MR spectroscopy of GABA levels in the anterior cingulate cortex
Resting state functional connectivity | Change from baseline to 1-week post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Leah Mayo, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No